CLINICAL TRIAL: NCT03197961
Title: The Pharmacokinetic and Pharmacodynamic Impacts of Depot Medroxyprogesterone Acetate on HIV Pre-exposure Prophylaxis (PrEP)
Brief Title: Pharmacokinetics and Pharmacodynamics of DMPA With HIV PrEP
Acronym: DynamoPrEP
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sharon Achilles (Other)
Responsible Party: Sponsor-Investigator, Sharon Achilles, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: PRO17010089
Record Dates: First submitted 2017-06-21; First posted 2017-06-23 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-12

CONDITIONS: HIV/AIDS; Contraception
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Tenofovir; Emtricitabine; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; N,N-dimethyl-4-anisidine; Medroxyprogesterone Acetate

STUDY DESIGN:
Intervention Model Description: This is a biphasic steady state pharmacokinetic and pharmacodynamic study of healthy women to evaluate the concentrations and activity of tenofovir and emtricitabine in different compartments before and after the administration of DMPA. Each participant will receive the study medications in the same order, i.e. TDF/FTC alone for 14 days followed by TDF/FTC for 14 days after having received DMPA.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- DMPA with tenofovir/emtricitabine PrEP (Experimental): the drug combination of tenofovir disoproxil fumarate 300mg and emtricitabine 200mg which is known as Truvada® will be taken orally once daily for 14 days by all participants. Drug concentrations will be measured (blood sampling) and one dose of Depot medroxyprogesterone acetate (DMPA) 150mg will be administered to each participant as an intramuscular injection after the first course of tenofovir disoproxil fumarate/emtricitabine is completed. Then, a second round of the combination of tenofovir disoproxil fumarate 300mg and emtricitabine 200mg (Truvada®) will be taken orally once daily for 14 days by all participants.
  Interventions: Combination Product: tenofovir/emtricitabine; Drug: DMPA

INTERVENTIONS:
Combination Product: tenofovir/emtricitabine — At the enrollment visit, participants will be given a 14-day supply of tenofovir/emtricitabine 200mg/300mg to take once daily for 14 days. Drug concentrations will be measured as outlined in the outcomes section at the end of the two week period. The tenofovir/emtricitabine 200mg/300mg course will be repeated approximately 2 to 6 weeks later to allow washout of tenofovir/emtricitabine.
  Other Names: Truvada®
Drug: DMPA — After completion of the first 14 day course of tenofovir/emtricitabine depot medroxyprogesterone acetate 150 mg will be administered as intramuscular injection.
  Other Names: Depot-Medroxyprogestereone Acetate

SUMMARY:
This study is a biphasic steady state pharmacokinetic and pharmacodynamic study of TFV and FTC in healthy women comparing the drug levels and activity in the absence (first phase) and then the presence (second phase) of DMPA. The investigators will recruit 12 healthy women aged 18-45 who are HIV-negative and at low risk for acquiring HIV.

DETAILED DESCRIPTION:
The investigators hypothesize that a drug interaction exists between DMPA and tenofovir/emtricitabine, such that levels of tenofovir (TFV) and emtricitabine (FTC) in cervicovaginal fluid, rectal fluid, and blood plasma, and levels of the active metabolites of TFV and FTC in cervical tissue and peripheral blood mononuclear cells will be significantly lower when women are using DMPA than when they are using no hormonal contraception. The investigators secondarily hypothesize that ex vivo HIV replication will be less suppressed in cervical tissue and cervicovaginal fluid when women are using the co-formulated pre-exposure prophylaxis oral pill containing tenofovir disoproxil fumarate (TDF), the prodrug of tenofovir, and FTC concurrently with the contraceptive injection DMPA as compared to when they are on TDF/FTC alone. This study is a biphasic steady state pharmacokinetic and pharmacodynamic study of TFV and FTC in healthy women comparing the drug levels and activity in the absence (first phase) and then the presence (second phase) of DMPA. The investigators will recruit 12 healthy women aged 18-45 who are HIV-negative and at low risk for acquiring HIV. Participants will take TDF/FTC for 14 days, after which drug levels will be measured and DMPA administered. After at least a 2 week washout period for TDF/FTC, participants will again take TDF/FTC for 14 days, and drug levels will be measured again. HIV replication activity will also be measured in cervicovaginal fluid and cervical tissue at baseline before starting TDF/FTC, after 14 days of TDF/FTC, and then after the second 14 days of TDF/FTC in the presence of DMPA.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-45 at screening
* In general good health and without any clinically significant systemic disease by history and per investigator judgement
* HIV negative at screening
* Heterosexually abstinent, consistent use of condoms, or female or male partner sterilization
* Currently having regular menstrual cycles (defined as cycles lasting 21-35 days by participant report)
* Agree not to participate in any other clinical trials involving drugs or medical devices during the study period
* Willing to comply with the study protocol

Exclusion Criteria:

* Currently or recently pregnant or breastfeeding (defined as pregnancy or breastfeeding in the last 3 months)
* Desiring pregnancy in the next 9 months
* Use of copper intrauterine device or other method of hormonal contraception
* Status post hysterectomy and/or bilateral oophorectomy
* Positive test for Hepatitis B surface antigen at screening
* Positive for Neisseria gonorrhea, Chlamydia trachomatis, or Trichomonas vaginalis at screening
* Positive syphilis screening test at screening
* Symptomatic bacterial vaginosis, defined as vaginal symptoms with Nugent score ≥ 7. (If symptomatic bacterial vaginosis is treated at screening and asymptomatic at enrollment, the participant may enroll.)
* Renal impairment (defined as creatinine clearance <60 ml/minute)
* Known bleeding disorder
* Daily use of NSAIDs
* Systemic use in the last two weeks or anticipated use during the study of any of the following: corticosteroids, antibiotics, anticoagulants, antifungals, antivirals, antiretrovirals, or other drugs known to prolong bleeding and/or clotting,
* Use of DMPA in the 6 months prior to screening
* Use of other hormonal contraception (including any contraceptive pill, patch, ring, implant, or levonorgestrel intrauterine device) in the 28 days prior to screening.
* Surgery requiring inpatient admission, or any abdominal surgery <30 days prior to enrollment
* Recreational or non-medical injection drug use in the 12 months prior to screening
* In a sexual relationship with a partner known to be HIV-positive or at high-risk of HIV (e.g. known recreational injection drug user, incarcerated in the 12 months prior to screening, etc.)
* Has any other condition that, in the opinion of the investigator, would preclude informed consent, make study participation unsafe, or complicate the interpretation of the study outcome data, or otherwise interfere with achieving the study objectives

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2017-11-17 (Actual); Primary Completion 2018-04-18 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Tenofovir and emtricitabine levels in the female genital tract, blood, and rectum | Two weeks after daily dosing of tenofovir/emtricitabine; before and after administration of depot medroxyprogesterone acetate
  The concentrations of tenofovir and emtricitabine in plasma, cervicovaginal fluid, and rectal fluid will be compared in women who are concomitantly using tenofovir/emtricitabine and DMPA as compared to using tenofovir/emtricitabine alone.

SECONDARY OUTCOMES:
Ex vivo HIV replication in cervical tissue and cervicovaginal fluid | Before tenofovir/emtricitabine and two weeks after daily dosing of tenofovir/emtricitabine both before and after administration of depot medroxyprogesterone acetate
  Ex vivo HIV replication in cervical tissue and cervicovaginal fluid will be compared in women who are concomitantly using tenofovir/emtricitabine and DMPA as compared to using tenofovir/emtricitabine alone

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Tarleton, MD, MPH, Principal Investigator — Clinical Instructor
Locations (1):
- Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No